CLINICAL TRIAL: NCT01027715
Title: The Impact of Electroencephalographic (EEG) Seizure Treatment in Near Term ≥ 36 Weeks Gestation and Term Infants With Neonatal Encephalopathy
Brief Title: The Impact of Electroencephalographic (EEG) Seizure Treatment in Neonatal Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-0888
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Seizures; Encephalopathy
Keywords: Neonatal Seizures; Neonatal encephalopathy
MeSH Terms: conditions — Seizures; Brain Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EEG seizure treatment group (Experimental): EEG data available to physicians. Treatment based on EEG seizures. Treatment will be dictated by the detailed treatment protocol. Standard antiepileptic medications will be used.
  Interventions: Other: EEG monitoring and treatment of EEG seizures
- Clinical Seizure treatment Group (No Intervention): Seizure treatment in this group will be based on standard care - treating clinical seizures only. While EEG data will be collected in this group, the data will not be available to the treating physicians. A one-hour EEG report will be available to the treating team. Continuous EEG monitoring and treatment will only be allowed if the initial EEG shows status.

INTERVENTIONS:
Other: EEG monitoring and treatment of EEG seizures — Seizures will prompt treatment with loading doses of phenobarbital (20mg/kg), fosphenytoin (20mg/kg),and midazolam (0.05mg/kg bolus and .15mg/kg/hr infusion tapered over 48 hours)in that order for persisting seizures.
  Other Names: EEG monitoring; Anti-epileptic drugs
  Arms: EEG seizure treatment group

SUMMARY:
This is a prospective, randomized, single-center pilot trial of term and near term (≥ 36 weeks gestation) infants with encephalopathy or seizures comparing a "EEG Seizure Treatment Group" or ESG with a "Clinical Seizure Treatment Group" or CSG.

The investigators hypothesize that the accurate detection and treatment of EEG seizures will decrease the seizure burden and improve outcomes in newborn infants with seizures and/or hypoxic-ischemic encephalopathy (HIE).

DETAILED DESCRIPTION:
This is a prospective, randomized, pilot trial of term and near term (≥ 36 weeks gestation) infants with encephalopathy or seizures comparing a "EEG Seizure Treatment Group" or ESG with a "Clinical Seizure Treatment Group" or CSG. Eligibility is based on clinical criteria for moderate/severe encephalopathy or seizures. We will recruit near term or term infants (≥ 36 weeks gestation) with a diagnosis of seizures or encephalopathy admitted to the neonatal intensive care unit (NICU) at St. Louis Children's Hospital within the first 72 hours of life. Infants will be randomized into an EEG Seizure Treatment Group (ESG) or a Clinical Seizure Treatment Group (CSG) (n=20 in each group). Patients in both groups will have EEG monitoring. While treating physicians will have access to EEG data in the ESG, no EEG data in the CSG will be available to the clinician for treatment of seizures. AED treatment will be initiated/escalated using stringent EEG seizure criteria (EST) or clinical criteria (CST) with the goal being seizure cessation. The specific AED, dosage, and duration of treatment is standardized in both groups. Monitoring will continue for a period of upto 96 hours in both arms. Other than the anticonvulsant drugs, treatment thresholds and dosing schedules, treatment in both arms will be at the discretion of the bedside physician.All infants will undergo an assessment of neuromotor disability and neurodevelopmental evaluation at 18 to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Term or near term infants ≥ 36 weeks gestation admitted to the neonatal intensive care unit
* ≤ 72 hours of age
* Screening for the "at risk" infant by the clinical team to include any one of the following:

  * Apgar score <5 at 5 min
  * Cord blood or postnatal gas with pH <7.0 or BE > -12
  * Need for respiratory support at 10 min of life
  * Suspected or definite seizures
  * Encephalopathy defined by recognition of altered neurological behavior
* Infants identified in the above screen will be examined by the research team and will be eligible if they satisfy at least one of the following:

  * Moderate-severe neonatal encephalopathy (3 out of 6 criteria)
  * Suspected or definite neonatal seizures

Exclusion criteria:

* Infants < 36 weeks gestation
* > 72 hours of age
* Infants with congenital anomalies of the central nervous system
* Moribund infants for whom no further aggressive treatment is planned
* Metabolic disorders or documented CNS infection
* Neuro-muscular blockade

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Seizure burden | 2 to 3 years
Presence of a single combined event: death in the first two years of life or moderate or severe disability at 18-24 months | first two years of life; 18-24 months

SECONDARY OUTCOMES:
Time to seizure cessation | 2 to 3 years
Number, duration of anticonvulsants used and cumulative dose | 2 to 3 years
EEG background state | 2 to 3 years
Time to all per oral feeding | 2 to 3 years
Duration of hospital stay | 2 to 3 years
MRI measures from the Day #7-10 MRI in survivors | 2 to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Mathur, Principal Investigator — Washington University in Saint Louis
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Srinivasakumar P, Zempel J, Trivedi S, Wallendorf M, Rao R, Smith B, Inder T, Mathur AM. Treating EEG Seizures in Hypoxic Ischemic Encephalopathy: A Randomized Controlled Trial. Pediatrics. 2015 Nov;136(5):e1302-9. doi: 10.1542/peds.2014-3777. Epub 2015 Oct 19. PMID 26482675